CLINICAL TRIAL: NCT02606994
Title: Comparison of the Healing of Chemotherapy-Induced Oral Mucositis Using Oral Defense Toothpaste Versus Crest Toothpaste and Magic Mouth Rinse
Brief Title: Effect of Over-the-counter Toothpastes on Chemotherapy-induced Oral Mucositis
Acronym: TPvsM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Oral Defense, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OralDefenseMucositisStudy
Record Dates: First submitted 2015-11-01; First posted 2015-11-17 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Mucositis; Neoplasms
Keywords: oral mucositis; chemotherapy; toothpaste
MeSH Terms: conditions — Mucositis; Neoplasms; Stomatitis | interventions — hydrated silica gel-based toothpaste; Lidocaine; aluminum hydroxide, magnesium hydroxide, drug combination; Diphenhydramine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Defense Toothpaste (Experimental): The experimental group will brush with Oral Defense Toothpaste three times per day during the study
  Interventions: Drug: Oral Defense Toothpaste
- Crest Toothpaste/Magic Mouth Rinse (Placebo Comparator): The placebo group will brush with Crest Toothpaste three times per day during the study. Participants in the placebo comparator group who require additional management of their oral mucositis pain will be provided Magic Mouth Rinse.
  Interventions: Drug: Crest Toothpaste; Drug: Magic Mouth Rinse

INTERVENTIONS:
Drug: Oral Defense Toothpaste — Brush with a Oral Defense Toothpaste three times per day during the study
  Other Names: Experimental toothpaste
  Arms: Oral Defense Toothpaste
Drug: Crest Toothpaste — Brush with Crest Toothpaste three times per day during the study
  Other Names: Control Toothpaste
  Arms: Crest Toothpaste/Magic Mouth Rinse
Drug: Magic Mouth Rinse — Participants using Crest Toothpaste who require additional pain intervention for their oral mucositis will be provided Magic Mouth Rinse
  Other Names: Viscous Lidocaine 2%, Maalox, Diphenhydramine 12.5mg/5ml
  Arms: Crest Toothpaste/Magic Mouth Rinse

SUMMARY:
The purpose of this study is to determine whether Oral Defense Toothpaste causes accelerated healing of chemotherapy-induced oral mucositis.

DETAILED DESCRIPTION:
A pilot study showed that patients with chemotherapy-induced oral mucositis experienced accelerated healing of their oral mucositis by brushing with Oral Defense Toothpaste.

In this study, participants experiencing up to grade 2 chemotherapy-induced oral mucositis will be split into two arms. The first arm (test arm) will receive Oral Defense Toothpaste and be required to brush three times per day, for 8 days. The second arm (control arm) will receive Crest Toothpaste and be required to brush three times per day, for 8 days. Patients in the control arm will be provided Magic Mouth Rinse, if needed. Healing of oral mucositis lesions will be evaluated at days 1 and 8. Quality of life assessment (determination of pain/loss of oral function) will be determined using a daily questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 receiving chemotherapy
* Mucositis lesions not exceeding grade 2

Exclusion Criteria:

* Patients receiving high load chemotherapy
* Patients receiving radiation therapy
* Patients receiving oral antivirals, oral antifungals or oral antibacterials
* Patients experiencing oral candidiasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Oral mucositis changes | Day 1 and 8 of the study
  The primary measure is the healing of chemotherapy induced oral mucositis lesions which are evaluated at days 1 and 8 of the study. The clinical investigators will identify patients who qualify for the study and this will mark day 1 of the study. At days 1 and 8 of the study, the clinical investigators will evaluate the oral cavity of each study participant and document changes in the oral mucositis of the participants.

SECONDARY OUTCOMES:
Quality of life changes | 8 days
  Each participant will fill out a quality of life questionnaire every day of the study. An evaluated outcome is when their chemotherapy induced oral mucositis lesions have resolved and their quality of life has returned to pre-chemotherapy levels.

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Chaudhry, MD,PhD, Principal Investigator — Summit Cancer Centers, Seattle Cancer Care Alliance
Locations (1):
- Summit Cancer Centers, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No